CLINICAL TRIAL: NCT02213913
Title: Prospective, Multi-center Phase I/II Trial of Lenalidomide and Dose-Adjusted EPOCH-R in MYC-Associated B-Cell Lymphomas
Brief Title: Lenalidomide and Combination Chemotherapy (DA-EPOCH-R) in Treating Patients With MYC-Associated B-Cell Lymphomas
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Chicago (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13-1406; NCI-2014-01581 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); IRB13-1406; 13-1406 (Other: University of Chicago); P30CA014599 (NIH)
Record Dates: First submitted 2014-08-05; First posted 2014-08-12 (Estimated); Last update posted 2023-04-28 (Actual); Status verified 2023-04

CONDITIONS: Adult Grade III Lymphomatoid Granulomatosis; B-cell Chronic Lymphocytic Leukemia; Contiguous Stage II Adult Diffuse Large Cell Lymphoma; Contiguous Stage II Adult Diffuse Mixed Cell Lymphoma; Contiguous Stage II Adult Diffuse Small Cleaved Cell Lymphoma; Contiguous Stage II Adult Immunoblastic Large Cell Lymphoma; Contiguous Stage II Grade 1 Follicular Lymphoma; Contiguous Stage II Grade 2 Follicular Lymphoma; Contiguous Stage II Grade 3 Follicular Lymphoma; Contiguous Stage II Mantle Cell Lymphoma; Contiguous Stage II Marginal Zone Lymphoma; Contiguous Stage II Small Lymphocytic Lymphoma; Cutaneous B-cell Non-Hodgkin Lymphoma; Extranodal Marginal Zone B-cell Lymphoma of Mucosa-associated Lymphoid Tissue; Intraocular Lymphoma; Nodal Marginal Zone B-cell Lymphoma; Noncontiguous Stage II Adult Diffuse Large Cell Lymphoma; Noncontiguous Stage II Adult Diffuse Mixed Cell Lymphoma; Noncontiguous Stage II Adult Diffuse Small Cleaved Cell Lymphoma; Noncontiguous Stage II Adult Immunoblastic Large Cell Lymphoma; Noncontiguous Stage II Grade 1 Follicular Lymphoma; Noncontiguous Stage II Grade 2 Follicular Lymphoma; Noncontiguous Stage II Grade 3 Follicular Lymphoma; Noncontiguous Stage II Mantle Cell Lymphoma; Noncontiguous Stage II Marginal Zone Lymphoma; Noncontiguous Stage II Small Lymphocytic Lymphoma; Progressive Hairy Cell Leukemia, Initial Treatment; Small Intestine Lymphoma; Splenic Marginal Zone Lymphoma; Stage 0 Chronic Lymphocytic Leukemia; Stage I Adult Diffuse Large Cell Lymphoma; Stage I Adult Diffuse Mixed Cell Lymphoma; Stage I Adult Diffuse Small Cleaved Cell Lymphoma; Stage I Adult Hodgkin Lymphoma; Stage I Adult Immunoblastic Large Cell Lymphoma; Stage I Chronic Lymphocytic Leukemia; Stage I Grade 1 Follicular Lymphoma; Stage I Grade 2 Follicular Lymphoma; Stage I Grade 3 Follicular Lymphoma; Stage I Mantle Cell Lymphoma; Stage I Marginal Zone Lymphoma; Stage I Small Lymphocytic Lymphoma; Stage II Adult Hodgkin Lymphoma; Stage II Chronic Lymphocytic Leukemia; Stage II Small Lymphocytic Lymphoma; Stage III Adult Diffuse Large Cell Lymphoma; Stage III Adult Diffuse Mixed Cell Lymphoma; Stage III Adult Diffuse Small Cleaved Cell Lymphoma; Stage III Adult Hodgkin Lymphoma; Stage III Adult Immunoblastic Large Cell Lymphoma; Stage III Chronic Lymphocytic Leukemia; Stage III Grade 1 Follicular Lymphoma; Stage III Grade 2 Follicular Lymphoma; Stage III Grade 3 Follicular Lymphoma; Stage III Mantle Cell Lymphoma; Stage III Marginal Zone Lymphoma; Stage III Small Lymphocytic Lymphoma; Stage IV Adult Diffuse Large Cell Lymphoma; Stage IV Adult Diffuse Mixed Cell Lymphoma; Stage IV Adult Diffuse Small Cleaved Cell Lymphoma; Stage IV Adult Hodgkin Lymphoma; Stage IV Adult Immunoblastic Large Cell Lymphoma; Stage IV Chronic Lymphocytic Leukemia; Stage IV Grade 1 Follicular Lymphoma; Stage IV Grade 2 Follicular Lymphoma; Stage IV Grade 3 Follicular Lymphoma; Stage IV Mantle Cell Lymphoma; Stage IV Marginal Zone Lymphoma; Stage IV Small Lymphocytic Lymphoma; Testicular Lymphoma; Untreated Hairy Cell Leukemia; Waldenström Macroglobulinemia
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Intraocular Lymphoma; Lymphoma, B-Cell, Marginal Zone; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Hodgkin Disease; Lymphoma, Large-Cell, Immunoblastic; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Waldenstrom Macroglobulinemia | interventions — Lenalidomide; Etoposide; Prednisone; Vincristine; Doxorubicin; Cyclophosphamide; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (lenalidomide, DA-EPOCH-R) (Experimental): INDUCTION PHASE: Patients receive lenalidomide PO daily on days 1-14. Treatment repeats every 21 days for 6 courses in the absence of disease progression or unacceptable toxicity.
  DA-EPOCH-R: Patients receive etoposide IV continuously on days 1-4, prednisone PO BID on days 1-5, vincristine sulfate IV continuously on days 1-4, doxorubicin hydrochloride IV continuously on days 1-4, cyclophosphamide IV over 15 minutes on day 5, and rituximab IV over 4 hours on day 1 (per institutional guidelines). Treatment repeats every 21 days for 6 courses in the absence of disease progression or unacceptable toxicity.
  CONSOLIDATION PHASE: Patients who are transplantation (HSCT)-eligible receive BEAM-conditioning regimen followed by autologous (auto)-HSCT or HSCT at the discretion of the treating physician. Patients who do not undergo HSCT in first remission receive lenalidomide maintenance for 12 months.
  Interventions: Drug: lenalidomide; Drug: etoposide; Drug: prednisone; Drug: vincristine sulfate; Drug: doxorubicin hydrochloride; Drug: cyclophosphamide; Biological: rituximab; Other: quality-of-life assessment; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: lenalidomide — Given PO
  Other Names: CC-5013; IMiD-1; Revlimid
Drug: etoposide — Given IV
  Other Names: EPEG; VP-16; VP-16-213
Drug: prednisone — Given PO
  Other Names: DeCortin; Deltra
Drug: vincristine sulfate — Given IV
  Other Names: leurocristine sulfate; VCR; Vincasar PFS
Drug: doxorubicin hydrochloride — Given IV
  Other Names: ADM; ADR; Adria; Adriamycin PFS; Adriamycin RDF
Drug: cyclophosphamide — Given IV
  Other Names: CPM; CTX; Cytoxan; Endoxan; Endoxana
Biological: rituximab — Given IV
  Other Names: IDEC-C2B8; IDEC-C2B8 monoclonal antibody; Mabthera; MOAB IDEC-C2B8; Rituxan
Other: quality-of-life assessment — Ancillary studies
  Other Names: quality of life assessment
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase I/II trial studies the side effects and best dose of lenalidomide when given together with combination chemotherapy and to see how well they work in treating patients with v-myc myelocytomatosis viral oncogene homolog (avian) (MYC)-associated B-cell lymphomas. Lenalidomide may stop the growth of B-cell lymphomas by blocking the growth of new blood vessels necessary for cancer growth and by blocking some of the enzymes needed for cell growth. Biological therapies, such as lenalidomide, use substances made from living organisms that may stimulate or suppress the immune system in different ways and stop cancer cells from growing. Drugs used in chemotherapy, such as etoposide, prednisone, vincristine sulfate, doxorubicin hydrochloride, cyclophosphamide, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Monoclonal antibodies, such as rituximab, may block cancer growth in different ways by targeting certain cells. Giving lenalidomide together with combination chemotherapy may be an effective treatment in patients with B-cell lymphoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the maximum tolerated dose (MTD) of lenalidomide when added to dose-adjusted (DA)-etoposide, prednisone, vincristine sulfate, doxorubicin hydrochloride, cyclophosphamide, rituximab (EPOCH-R) (hereby termed "DA-EPOCH-RR") in patients with double hit lymphoma (DHL) lymphomas. (Phase I) II. To determine the 1- and 2-year progression free survival (PFS) of DA-EPOCH-RR in patients with DHL lymphomas. (Phase II)

SECONDARY OBJECTIVES:

I. Overall response rate, complete response, and duration of response. II. Quality of life (QOL) measures using standardized scales. III. Toxicity assessment using version 4.0 of the National Cancer Institute (NCI)-Common Terminology Criteria for Adverse Events (CTCAE) criteria.

IV. Overall survival (OS) at 1 and 2 years.

OUTLINE: This is a phase I, dose-escalation study of lenalidomide followed by a phase II study.

INDUCTION PHASE: Patients receive lenalidomide orally (PO) daily on days 1-14. Treatment repeats every 21 days for 6 courses in the absence of disease progression or unacceptable toxicity.

DA-EPOCH-R: Patients receive etoposide intravenously (IV) continuously on days 1-4, prednisone PO twice daily (BID) on days 1-5, vincristine sulfate IV continuously on days 1-4, doxorubicin hydrochloride IV continuously on days 1-4, cyclophosphamide IV over 15 minutes on day 5, and rituximab IV over 4 hours on day 1 (per institutional guidelines). Treatment repeats every 21 days for 6 courses in the absence of disease progression or unacceptable toxicity.

CONSOLIDATION PHASE: Patients who are transplantation (hematopoietic stem cell transplant [HSCT])-eligible receive BCNU, etoposide, cytarabine, and melphalan (BEAM)-conditioning regimen followed by autologous (auto)-HSCT or HSCT at the discretion of the treating physician. Patients who do not undergo HSCT in first remission receive lenalidomide maintenance for 12 months.

After completion of study treatment, patients are followed up for every 3 months for 1 year, every 4 months for 1 year, and then periodically for 1 year.

ELIGIBILITY:
Inclusion Criteria

1. B-cell lymphoma with comprehensive immunohistochemistry (IHC) panel establishing lineage (CD20, CD3) and cell of origin (CD10, BCL6 and MUM1) in addition to proliferative/prognostic markers (Ki-67, C-myc and BCL2). DHL will be identified using cytogenetics and/or immunohistochemistry as detailed in section 4.1.2 below.
2. To define DHL, patients must have evidence of C-myc [defined as: Cytogenetic evidence (FISH or karyotype) of C-myc breaks (Increased copy number in itself is not considered positivity for C-myc) OR Positive IHC defined as >40% of the lymphoma cells staining for C-myc] PLUS either:

   1. Breaks in BCL-2 via cytogenetic studies or
   2. BCL-2 immunopositivity in >70% of lymphoma cells.
3. Patients are allowed to have received radiotherapy before enrollment if radiation was given to alleviate pain and/or neurologic compromise as long as there remains areas of measurable disease present. Further, at the investigator's discretion and for patients who are unstable, one cycle of R-CHOP is allowed prior to enrollment but no more than one cycle. For purposes of this trial, prednisone or other corticosteroids used for non-lymphomatous conditions will be allowed. In addition, a prior/recent short course (< 2 weeks) of steroids for symptom relief of lymphoma-related symptoms will be allowed.
4. AST and ALT < 3 x upper limit of normal (ULN), and total bilirubin <1.5 x ULN (with exception of patients with Gilbert's syndrome, asymptomatic gallstones, liver involvement with NHL or stable chronic liver disease per investigator assessment).
5. Patients must have adequate renal function by virtue of GFR > 50 ml/minute using Cockroft-Gault formula.
6. Patients must have adequate bone marrow function (platelets >100,000 and ANC >1,200). Patients with bone marrow involvement are allowed at the investigator's discretion regardless of cytopenias.
7. ECOG PS 0-2.
8. Age ≥ 18 years.
9. All study participants must be registered into the mandatory lenalidomide REMS® program, and be willing and able to comply with the requirements of the REMS® program.
10. Females of reproductive potential must adhere to the scheduled pregnancy testing as required in the lenalidomide REMS® program. (Please see study schema for further details)
11. Able to take aspirin (81 or 325 mg) daily as prophylactic anticoagulation (patients intolerant to ASA may use warfarin or low molecular weight heparin).
12. Ability to read, understand, and sign a written informed consent approved by each institutional IRB. Alternatively, patients with legal guardians who can read, understand, and sign written informed consent may also enroll.

Exclusion Criteria

1. Prior therapy for lymphoma
2. Known CNS involvement
3. Known HIV positive status
4. Pregnant females
5. Burkitt and/or precursor lymphoblastic leukemia/lymphoma.
6. Prior pomalidomide exposure
7. Known hypersensitivity to lenalidomide or thalidomide
8. The development of erythema nodosum if characterized by a desquamating rash while taking thalidomide or similar drugs.
9. Subjects who have currently active hepatic or biliary disease (with exception of patients with Gilbert's syndrome, asymptomatic gallstones, liver involvement with NHL or stable chronic liver disease per investigator assessment).
10. Treatment with any known non-marketed drug substance or experimental therapy within 4 weeks prior to enrollment, or currently participating in any other interventional clinical study for NHL or any other illness (except observational, prevention, and/or registry trials).
11. No current malignancy. Subjects who have been free of malignancy for at least 2 years, or have a history of completely resected non-melanoma skin cancer, or successfully treated in situ carcinoma (any site) are eligible. Women with a history of cervical cancers are allowed.
12. Chronic or current infectious disease requiring systemic antibiotics, antifungal, or antiviral treatment such as, but not limited to, chronic renal infection, chronic chest infection with bronchiectasis, tuberculosis and active Hepatitis C.
13. History of significant cerebrovascular disease in the past 3 months or ongoing event with active symptoms or sequelae.
14. Positive serology for Hepatitis B (HB) defined as a positive test for HBsAg. In addition, if negative for HBsAg but HBcAb positive (regardless of HBsAb status), a HB DNA test will be performed and if positive, the subject will be excluded if unable to tolerate and/or receive anti-Hepatitis-B therapy. Positive serology because of prior vaccination is allowed.
15. Positive serology for hepatitis C (HC) defined as a positive test for HCAb.
16. Inability to comply with study or follow-up testing and procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2014-07-29 (Actual); Primary Completion 2023-07-29 (Estimated); Study Completion 2023-07-29 (Estimated)

PRIMARY OUTCOMES:
PFS | Time elapsed between treatment initiation and tumor progression or death from any cause (whichever occurs first), assessed up to 3 years
MTD of adding lenalidomide to the DA-EPOCH-R regimen as a front-line therapy in patients with DHL lymphomas (using CTCAE v 4.0) (Phase I) | Up to 21 days
PFS (Phase II) | Time elapsed between treatment initiation and tumor progression or death from any cause (whichever occurs first), assessed at 1 year
PFS (Phase II) | Time elapsed between treatment initiation and tumor progression or death from any cause (whichever occurs first), assessed at 2 years

SECONDARY OUTCOMES:
Add lenalidomide to the DA-EPOCH-R regimen as a front-line therapy in patients with DHL lymphomas (Phase I) | Up to 18 weeks
  Time elapsed between treatment initiation and tumor progression or death from any cause (whichever occurs first), assessed up to 18 weeks
Overall response rate defined as the sum of partial response (PR) and complete response (CR) by computed tomography (CT) of positron emission tomography/CT and/or resolution of marrow-only involvement (if originally involved) (Phase I) | Up to 18 weeks
Anti-tumor activity, calculated as the sum of stable disease, PR, and CR according to the Revised Response Criteria for Malignant Lymphoma and Cheson et al (Phase I) | Up to 18 weeks
Duration of response, calculated as the duration from detecting any objective response until progression or death from any cause, according to the Revised Response Criteria for Malignant Lymphoma and Cheson et al (Phase I) | Time elapsed between initial documented PR or CR and first progression event, assessed up to 18 weeks
Incidence of adverse events, defined as the occurrence of all grades of toxicity (using CTCAE version 4.0) | Up to 21 days from last treatment
  The occurrence and severity of each event will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Sonali Smith, Principal Investigator — University of Chicago
Locations (6):
- United States (6):
  - Rush University Medical Center, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - Decatur Memorial Hospital Cancer Care Institute, Decatur, Illinois
  - NorthShore University HealthSystem, Evanston, Illinois
  - Illinois Cancer Care, Peoria, Illinois
  - University of Maryland, Baltimore, Maryland

REFERENCES:
- [Derived] Cahill K, Godfrey J, Nabhan C, Kline J, Riedell PA, Cohen KS, Narula S, Karrison TG, Robertson J, Karmali R, Venugopal P, Kim SH, Rapoport AP, Lee ST, Law J, Fishkin PAS, Isufi I, Velasco M, Kaminer L, Smith SM. A multicenter phase 1/2 trial of lenalidomide and dose-adjusted EPOCH-R in MYC-associated DLBCL. Blood Adv. 2025 Nov 11;9(21):5665-5675. doi: 10.1182/bloodadvances.2025017092. PMID 40720747